CLINICAL TRIAL: NCT04070898
Title: Prospective, Controlled, Randomized Multicentric Study of Non-inferiority on the Management of the Vesical Catheter in Colon Surgery. CR-Vesical Cath Study Group
Brief Title: Prospective, Controlled, Randomized Multicentric Study on the Management of the Vesical Catheter in Colon Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Principal Investigator, Head Colorectal Unit, Clinical Professor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-Vesical Cath-2019-01
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Colon Cancer
Keywords: Laparoscopic colectomy; urinary catheter; acute urinary retention
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: A multicenter prospective, controlled, randomized, non-inferiority study on the management of the bladder catheter in scheduled laparoscopic colon surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Bladder catheter removal 24 hours after surgery
- experimental group (Experimental): Removal of the bladder catheter after the surgical intervention
  Interventions: Procedure: Remove urinary catheter after surgery

INTERVENTIONS:
Procedure: Remove urinary catheter after surgery — Remove bladder catheter after surgery
  Arms: experimental group

SUMMARY:
INTRODUCTION: Recommendations for peroperative bladder catheterization remain a controversial issue since it is a procedure that is not without complications. Most of the current suggestions derive from open surgery data that have been extrapolated to Enhanced Recovery After Surgery (ERAS) or Fast-Track programs ranging between 24-48 hours.

The objective of the present study is to find the perfect balance with a better degree of evidence than the current one between the reduction of the probing time and the non-increase of the acute retention of urine in the patients operated in a programmed way of laparoscopic colon surgery.

Methods: Multicenter, prospective, controlled, randomized non-inferiority study on the management of the bladder catheter in patients undergoing scheduled laparoscopic colon surgery, randomized in two study groups: experimental group (removal of the bladder catheter after surgery ) and control group (removal of the catheter at 24 hours) after the surgical intervention.

The main objective of the present study is to reduce the permanence of the bladder catheter trying to find the balance of the probing time and the non-increase of the acute retention of urine in the patients operated in a programmed way of laparoscopic colon surgery As secondary objectives we will consider the decrease in the incidence of urinary tract infections within the first 30 days as well as the reduction in hospital stay and morbidity related to the bladder catheter.

DETAILED DESCRIPTION:
INTRODUCTION: The usual recommendations for a peroperative bladder catheter vary from surgical reasons to the control of hemodynamics or personal preferences, so since it is not a procedure free of complications, it requires an evidence-based approach.

For hospitalized patients, the optimal duration of bladder catheterization remains controversial. For colorectal surgery, most authors traditionally suggested with limited evidence, based mainly on open surgery data, 5 days with a range of 3 to 10 days, which meant a significant increase in hospital stays associated with an increase of the risk of complications (42-60% of urinary infections).

With the introduction of the Enhanced Recovery After Surgery (ERAS) or Fast-Track programs of minimally invasive surgery it has been shown that old concepts adopted by the inertia of the custom were wrong and therefore the recommended duration of bladder catheterization has been shortened with the aim of reducing the incidence of urinary tract infections without significantly increasing acute urinary retention.

Currently, European international guidelines recommend that bladder catheterization may be limited to a period of 24-48 hours after scheduled colon and rectal interventions, except for resections of the middle and lower rectum (with extensive perineal and rectal dissection) that require the permanence of the bladder catheter for a longer period according to the clinical indications.

The clinical guidelines of the ASCRS (American Society of Colon and Rectal Surgeons) and the SAGES (Society of American Gastrointestinal and Endoscopic Surgeons) are even more restrictive in the use of bladder catheterization in elective colon or upper rectum surgery, recommending its withdrawal within 24 hours after it as they consider that at 48 hours the risk of postoperative urinary tract infection has doubled.

HYPOTHESES AND OBJECTIVES Hypothesis: Although the ERAS guidelines recommend the removal of the bladder catheter at 24 hours or 2-3 days, we believe that it can be removed earlier at the end of surgery without detriment to the increase in acute retention of urine and with the benefit of earlier mobilization and decreased morbidity related to the bladder catheter (urine infection).

The main objective of the study is the assessment of the degree of acute retention of urine after removal of the bladder catheter in colon surgery in the two study groups, control (24 h) and in the experimental group (once the surgical intervention ends ).

As secondary objectives we will consider the decrease in the incidence of urinary tract infections within the first 30 days as well as the reduction in hospital stay and morbidity related to the bladder catheter. Urine culture samples will be collected if the patient presents a clinic suggestive of urinary tract infection: dysuria, urinary frequency, urgency, suprapubic pain, hematuria or testicular pain.

METHODS / DESIGN Study design This protocol has been designed following the standards of the SPIRIT statement and is a prospective, multicentre, controlled, randomized, non-inferiority study on the management of the bladder catheter in scheduled laparoscopic colon surgery

Inclusion criteria Any patient who understands, agrees to participate and signs the informed consent, that is over 18 years old, operated electively and programmed by laparoscopic colon and upper rectum in which the peritoneal reflection has not been opened, will be included in the study. with a duration of the surgical act less than 180 minutes. The previous anesthetic assessment will be of an ASA I-III and should have an international prostate symptom score (IPSS) of less than 19 with / without treatment for BPH (alpha-blocker).

Exclusion criteria Open surgery or conversion to open surgery; performing periodic anesthesia or being ASA IV; preoperative diagnosis of urinary tract infections (more than 3 episodes / year documented by urinoculture or two urinary tract infections in the last 6 months); moderate-severe prostate clinic (IPSS> 19); in men, the presence of positive urine culture in preoperative tests; in women, the urinary infection clinic and the positive urine culture. The previous history of acute urine retention will also be grounds for exclusion from the study; be a carrier of a permanent bladder catheter or ureteral catheter and intermittent self-catheterization. Men who have undergone prostatic deobstructive surgery (Holep, RTUp, Millin or prostatic vaporization) will not be included; patients with a history of treatment for urological tumor (prostate cancer, bladder tumor, ureteral or renal tumor); or have a history of urethral stricture, enterovesical fistula or previous pelvic surgery. Other reasons for exclusion will be urinary incontinence or neurogenic bladder; chronic renal failure (CRF) with creatinine levels greater than 2 (including terminal CRI stage or dialysis); emergency surgery, pregnant women, having received pelvic radiotherapy or the administration of suerotherapy during the operative time> 2,000ml.

Study withdrawal criteria The difficulty / impossibility of intraoperative catheterization, urethral bleeding / hematuria after traumatic catheterization or the need for suprapubic cystostomy placement; the patient who is under active antibiotic treatment due to urinary tract infection at the time of surgery; the need for intraoperative ureteral catheter placement; the need for 24-hour diuresis monitoring by bladder catheterization, the combination with other surgeries (hysterectomy, prostatectomy, etc.), Clavien post-surgical complications> 2 (need to take a probe longer than expected); intraoperative urinary tract injury or the need for peridural anesthesia in the immediate postoperative period.

The preoperative evaluation in men will include an IPSS questionnaire and a urine culture as its positivity will mean exclusion from the study. It will also be evaluated if you take medication for BPH. In women, a urine culture will be performed in case of presenting a urinary infection clinic

Recruitment and scope of the study Patients will be recruited from colorectal surgery units of hospitals participating in the study following the same criteria.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who understands, agrees to participate and signs the informed consent
* older than 18 years-old
* electively operated and programmed laparoscopically of the colon and upper rectum in which peritoneal reflection has not been opened
* duration of the surgical act less than 180 minutes
* Prior anesthetic assessment of ASA I-III
* International prostate symptom score (IPSS) of less than 19 with / without treatment for BPH (alpha-blocker).

Exclusion Criteria:

* - Open surgery or conversion to open surgery
* Performing periodic anesthesia or being ASA IV
* Preoperative diagnosis of recurrent urinary tract infections (more than 3 episodes / year documented by urinoculture or two urinary tract infections in the last 6 months);
* Moderate-severe prostate clinic (IPSS> 19)
* Presence of positive urine culture in men in preoperative tests
* Urinary infection clinic in women with positive urine culture
* Previous history of acute urine retention
* be a permanent bladder catheter or ureteral catheter and perform intermittent autocatheterization.
* men who underwent prostate surgery
* patients with a history of treatment for urological tumor - patients with a history of urethral stricture, enterovesical fistula or previous pelvic surgery.
* urinary incontinence or neurogenic bladder
* chronic renal failure (CRF) with creatinine levels greater than 2 (including terminal CRI stage or dialysis)
* emergency surgery pregnant
* have received pelvic radiotherapy
* Administration of serum during the operative time> 2,000ml.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of acute urine retention after removal of the bladder catheter after colon surgery. | 8 hours
  Acute urine retention is defined as
  * the inability to spontaneous urination at 8 hours after the removal of the bladder catheter
  * obtaining after urinary catheterization of more than 400 cc of urine or the need for repeated probing due to the impossibility of spontaneous urination

SECONDARY OUTCOMES:
Change incidence of urinary tract infections | 30 days
  Urine culture is more than 10,000 colonies per ml in men or 100,000 colonies per ml in women produced by 1 or 2 microorganisms.
Change of hospital stay | 30 days
  hospital stay less than usual in this surgery
Morbidity changes | 30 days
  According to the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD, PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Hospital Universitario Parc Tauli de Sabadell, Sabadell, Barcelona, Spain